CLINICAL TRIAL: NCT02974283
Title: The Effect of Normobaric Hyperoxia on Blood Brain Barrier in AIS Patients Based on a Blood Marker for the Evaluation of Blood Brain Barrier Damage From Animal Experiments
Brief Title: Protective Effects of Normobaric Hyperoxia on Blood Brain Barrier in Patients With Acute Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming, professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBO-2016
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Stroke, Acute
Keywords: Normobaric hyperoxia; r-tPA thrombolytic therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NBO group (Experimental): Normobaric oxygen therapy is the delivery of high-flow oxygen (10L/min) via oxygen storage facemask. This therapy should start within 1 hours after diagnosis of ischemic stroke and last for 4hours. All participants will receive r-tPA thrombolytic therapy and a standard clinical therapy.
  Interventions: Other: Normobaric oxygen therapy
- Control group (No Intervention): The participants receive r-tPA thrombolytic therapy after diagnosed ischemic. All participants receive a standard clinical therapy.

INTERVENTIONS:
Other: Normobaric oxygen therapy — In this study, it is simple to administer via oxygen storage facemask at flow rates of 10 L/min for 4 hours. This therapy start should within 1 hour after diagnosed ischemic stroke and uninterrupted during other treatments including r-tPA thrombolytic therapy and standard clinical treatment. .
  Other Names:
  Arms: NBO group

SUMMARY:
The purpose of this study is to find out a serum marker for the evaluation of blood brain barrier damage based on animal experiments and investigate the effect of NBO（Normobaric hyperoxia）on blood brain barrier in the acute ischemic stroke patients who received r-tPA thrombolytic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female with age from 18 to 85;
2. Acute ischemic stroke;
3. National Institutes of Health Stroke Scale (NIHSS) score of 4-25
4. mRS score less than 1 before onset of stroke symptom;
5. Onset of stroke symptoms within 4.5h before initiation of intravenous r-tPA thrombolytic therapy;
6. Informed consent obtained

Exclusion Criteria:

1. Stroke or serious head trauma within the previous 3 months
2. Major surgery or severe trauma with in the preceding 3 months
3. Intracranial hemorrhage
4. Systolic pressure greater than 185 mm Hg or diastolic pressure greater than 110 mm Hg, or aggressive treatment intravenous medication) necessary to reduce blood pressure to these limits
5. Symptoms rapidly improving
6. Symptoms suggestive of subarachnoid hemorrhage, even if CT scan was normal
7. Gastrointestinal hemorrhage or urinary tract hemorrhage within the previous 21 days
8. Arterial puncture at a noncompressible site within the previous 7 days
9. Seizure at the onset of stroke
10. Platelet count of less than 100,000 per cubic millimeter
11. Received heparin within the 48 hours preceding the onset of stroke and had an elevated partial-thromboplastin time
12. Received oral anticoagulation therapy preceding the onset of stroke and INR greater than 1.7 or prothrombin times greater than 15 seconds
13. CT showed a multiple infarction (low density area greater than 1/3 cerebral hemisphere)
14. severe hepatic or renal dysfunction
15. active and chronic obstructive pulmonary disease or acute respiratory distress syndrome;
16. >3 L/min oxygen required to maintain peripheral arterial oxygen saturation (SaO2)﹥95% as per current stroke management guidelines; 17 medically unstable;

18. inability to obtain informed consent. 19. Life expectancy<1 years 20. Pregnant or breast-feeding women 21. Unwilling to be followed up or poor compliance for treatment 22. Patients being enrolled or having been enrolled in other clinical trial within 3 months prior to this clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
levels of blood biomarkers | 7days
  a serum marker for the evaluation of blood brain barrier damage based on animal experiments
Scores assessed by National Institutes of Health Stroke Scale(NIHSS) | 7days

SECONDARY OUTCOMES:
Number of participants with adverse events that are related to treatment | 7days

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD. Ph.D, Principal Investigator — Capital Medical University

REFERENCES:
- [Derived] Shi S, Qi Z, Ma Q, Pan R, Timmins GS, Zhao Y, Shi W, Zhang Y, Ji X, Liu KJ. Normobaric Hyperoxia Reduces Blood Occludin Fragments in Rats and Patients With Acute Ischemic Stroke. Stroke. 2017 Oct;48(10):2848-2854. doi: 10.1161/STROKEAHA.117.017713. Epub 2017 Sep 20. PMID 28931617